CLINICAL TRIAL: NCT04603924
Title: A Phase 2/3 Randomized and Placebo-Controlled Study of ANA001 in Moderate and Severe COVID-19 Patients
Brief Title: Study of Niclosamide in Moderate and Severe Hospitalized Coronavirus-19 (COVID-19) Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANA001-001
Record Dates: First submitted 2020-10-20; First posted 2020-10-27 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
Keywords: Corona Virus Disease (COVID-19); Niclosamide; Antiviral; Immunomodulator; Oral Niclosamide; Infection; Acute Respiratory Distress Syndrome (ARDS); Cytokine dysregulation; Virus; Viral; anthelmintic; anti-inflammatory; bronchodilator; antineoplastic; ANA001; Moderate COVID-19; ARDS; Acute Respiratory Distress Syndrome; Hospitalized COVID-19
MeSH Terms: conditions — COVID-19; Infections; Respiratory Distress Syndrome; Virus Diseases | interventions — Niclosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ANA001 (Experimental): Subjects in the ANA001 treatment arm will receive 1,000 mg (4 capsules; 250 mg each) by mouth twice per day for 7 consecutive days with a meal. If the participant requires mechanical ventilation over the course of the study, ANA001 may be administered via nasogastric (NG), percutaneous endoscopic gastrostomy (PEG) or orogastric (OG) tube and, if possible, should be administered with a scheduled nasogastric (NG) or orogastric (OG) feeding.
  Interventions: Drug: Niclosamide
- Matching Placebo (Placebo Comparator): Subjects in the comparator arm will receive matching placebo (hydroxypropylmethylcellulose (HPMC)) (4 capsules, by mouth twice a day) for the 7-day treatment duration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niclosamide — Niclosamide is an antihelmintic with in-vitro antiviral activity
  Other Names: ANA001
  Arms: ANA001
Drug: Placebo — Matching hydroxypropylmethylcellulose HPMC capsules with no active ingredients
  Other Names: Matching Placebo to ANA001
  Arms: Matching Placebo

SUMMARY:
Study of ANA001 in Moderate and Severe COVID-19 Patients

DETAILED DESCRIPTION:
This is a 2 part, Phase 2/3 multi-center, double blinded, placebo-controlled study to assess the safety, tolerability, and efficacy of oral niclosamide (ANA001) in moderate and severe hospitalized COVID-19 patients compared to placebo.

ELIGIBILITY:
Key Inclusion Criteria:

1. Provide written informed consent prior to performing study procedures
2. Hospitalized.
3. Male or female ≥18 years of age
4. Positive for severe acute respiratory syndrome coronavirus 2
5. Presence of symptoms of lower respiratory tract infection (LRTI) including at least 1 of the following: fever, cough, sore throat, malaise, headache, muscle pain, or more significant lower respiratory tract symptoms, including shortness of breath
6. At least 1 of the following: respiratory rate (RR) ≥20 breaths per minute, room air oxygen saturation (SpO2) <98%, requirement for supplemental oxygen, heart rate (HR) ≥90 beats per minute, or temperature >38.3°C
7. Women of childbearing potential must agree to abstinent or use at least 1 form of contraception not including hormonal contraception from the day of screening through Day 30

Key Exclusion Criteria:

1. Hospitalized but no longer requires ongoing inpatient care (i.e., discharge is anticipated in ≤24 hours)
2. Patient is not anticipated to survive >48 hours OR is under palliative care
3. Evidence of critical illness, defined by at least 1 of the following:

   * Respiratory failure requiring at least 1 of the following:

     1. Endotracheal intubation and mechanical ventilation, oxygen delivered by high flow nasal cannula
     2. Noninvasive positive pressure ventilation (NIPVV), OR
     3. Extracorporeal membrane oxygenation (ECMO) or clinical diagnosis of respiratory failure
   * Shock (defined by systolic blood pressure (BP) <90 mm Hg, or diastolic blood pressure (BP) <60 mm Hg or requiring vasopressors), OR
   * Multi-organ dysfunction/failure
4. Severe central nervous system (CNS) conditions
5. Chronic kidney disease requiring dialysis
6. Known allergy to the study drug or salicylate containing medications.
7. Suspected and/or confirmed pregnancy or breastfeeding
8. Current or planned participation in any other clinical trial of a treatment being developed under a US investigational new drug (IND) or emergency use authorization (EUA).
9. Patients receiving chemotherapeutic agents and/or immunomodulators (including monoclonal antibodies (Mabs) or plasma transfusions) for chronic disease conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doug Rank, MD, Study Director — NeuroBo Pharmaceuticals
Locations (8):
- United States (8):
  - Helen Keller Hospital, Sheffield, Alabama
  - University of California, Irvine, Irvine, California
  - Baptist Health Research Institute, Jacksonville, Florida
  - AdventHealth Tampa, Tampa, Florida
  - University of Missouri Health Care, Columbia, Missouri
  - Caroline Institute for Clinical Research, Fayetteville, North Carolina
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - Providence Regional Medical Center Everett, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ANA001 | Matching Placebo
Started | 25 | 24
Subjects Dosed | 23 (2 randomized subjects withdrew/ were withdrawn prior to dosing. 1 further subject (102015) withdrew consent after receiving 1 dose of Active Treatment (ANA001). This subject was not included in either Pharmacokinetic (PK) or Safety analysis sets.) | 23 (1 randomized subject withdrew/ was withdrawn prior to dosing.)
Completed | 15 | 15
Not Completed | 10 | 9
Not completed — Not Dosed | 2 | 1
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ANA001 | Matching Placebo | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Customized [Count of Participants; unit: Participants]
  18 -<40 Years | 5 | 3 | 8
  40-<65 Years | 13 | 15 | 28
  >/=65 Years | 7 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 12 | 14 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 17 | 18 | 35
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 20 | 18 | 38
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Days from First COVID-19 Symptom to Randomisation [Mean (Standard Deviation); unit: Days] — Date of Randomization minus the Date of the first COVID-19 symptom
  Days | 7.6 (4.12) | 7.7 (3.53) | 7.7 (3.81)
Baseline WHO Ordinal Scale for Clinical Improvement [Count of Participants; unit: Participants] — This is a 9 point ordinal scale with 0 indicating "No clinical or virological evidence of infection" and 8 indicating "Death".
  Participants
    Baseline World Health Organisation (WHO) Ordinal Scale for Clinical Improvement= 4 | 3 | 4 | 7
    Baseline World Health Organisation (WHO) Ordinal Scale for Clinical Improvement = 5 | 19 | 17 | 36
    Baseline World Health Organisation (WHO) Ordinal Scale for Clinical Improvement = 6 | 1 | 2 | 3
    Baseline World Health Organisation (WHO) Ordinal Scale for Clinical Improvement = Missing | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing TEAEs
Description: Incidence of Treatment Emergent Adverse Events (TEAEs)
Time Frame: Randomization to Day 60
Population: Safety Analysis Set: Includes all randomized participants, classified according to the actual treatment received regardless of randomization assignment, who received any amount of study drug and have at least one post-baseline safety evaluation. This is the analysis population for all planned safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | ANA001 | Matching Placebo
Number analyzed (Participants) | 22 | 23
Participants
  No. of Subjects with any TEAE | 16 | 12
  No. of Subjects with Mild (Grade 1) TEAEs | 9 | 2
  No. of Subjects with Moderate (Grade 2) TEAEs | 5 | 4
  No. of Subjects with Severe (Grade 3) TEAEs | 0 | 2
  No. of Subjects with Life-Threatening (Grade 4) TEAEs | 0 | 1
  No. of Subjects with Death (Grade 5) TEAEs | 2 | 3

2. Primary Outcome: Number of Subjects Experiencing TESAEs
Description: Incidence of Treatment Emergent Serious Adverse Events (TESAEs)
Time Frame: Randomization to Day 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ANA001 | Matching Placebo
Number analyzed (Participants) | 22 | 23
Participants | 3 | 6

3. Secondary Outcome: Median Time to Hospital Discharge
Description: Median time until patient is discharged from hospital. Discharge is defined as a score of 1 or 2 in the WHO Ordinal Scale for Clinical Improvement. This is a 9 point ordinal scale with 0 indicating "No clinical or virological evidence of infection" and 8 indicating "Death".
Time Frame: Randomization to Day 60
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ANA001 | Matching Placebo
Number analyzed (Participants) | 23 | 23
Days | 6.03 [3.07 to 14.89] | 13.92 [5.85 to NA] — Median time to hospital discharge and corresponding 95% C.I. were estimated from the Kaplan-Meier curves. In some cases the 95% confidence interval could not be calculated due primarily to censoring of data: Participants who are lost to follow-up as of the data analysis cutoff date are censored on the date of the participant's last known WHO Ordinal Scale for Clinical Improvement; Participants who die in the hospital are right censored at Day 60 or date of death, whichever is earlier.
Statistical Analysis 1: Comparison: ANA001 vs Matching Placebo; Test type: Other; For the analysis of this efficacy endpoint, missing scores of the WHO Ordinal Scale for Clinical Improvement will be assumed to be > 2 (i.e., no hospital discharge). Median time-to-clinical improvement and corresponding 95% confidence interval were estimated from the Kaplan-Meier curves. In some cases the 95% confidence interval was "Not Evaluable" (NE) by this method

4. Secondary Outcome: Median Time to 2-point Improvement WHO Clinical Improvement Scale
Description: Median Time to 2-point Improvement in WHO Ordinal Scale for Clinical Improvement. This is a 9 point ordinal scale with 0 indicating "No clinical or virological evidence of infection" and 8 indicating "Death"
Time Frame: Randomization to Day 60
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | ANA001 | Matching Placebo
Number analyzed (Participants) | 23 | 23
Days | 4.15 [2.98 to 6.96] | 13.91 [5.85 to NA] — Median Time to 2-point Improvement in WHO Ordinal Scale for Clinical Improvement and corresponding 95% confidence interval were estimated from the Kaplan-Meier curves. In some cases the 95% confidence interval could not be calculated by this method primarily due to data censoring: participants lost to follow up are censored on the date of the participant's last known WHO Ordinal Scale for Clinical Improvement. Participants who die in the hospital are right censored at Day 60.
Statistical Analysis 1: Comparison: ANA001 vs Matching Placebo; Test type: Other; For the analysis of this efficacy endpoint, missing scores of the WHO Ordinal Scale for Clinical Improvement were be assumed to be > 2 (i.e., no hospital discharge). Median number of days to a 2-point improvement and corresponding 95% confidence interval were estimated from the Kaplan-Meier curves. In some cases the 95% confidence interval was "Not Evaluable" (NE) by this method

5. Secondary Outcome: Median Time to Resolution of COVID-19 Symptoms
Description: Median time (in days) to resolution of subjective symptoms assessed by the Investigator to be potentially due to COVID-19 including: fever, cough (productive or non-productive), sore throat, malaise, headache, muscle pain, gastrointestinal symptoms (i.e., nausea, vomiting, or diarrhea), shortness of breath (with or without exertion), and respiratory distress
Time Frame: Randomization to Day 60
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ANA001 | Matching Placebo
Number analyzed (Participants) | 23 | 23
Days | 17 [9 to 36] | 16 [11 to 24]

6. Secondary Outcome: Median Time to Time-to-Viral Load Undetectable
Description: Median number of days to viral load undetectable by nasopharyngeal (NP) swab
Time Frame: Randomization to Day 60
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ANA001 | Matching Placebo
Number analyzed (Participants) | 23 | 23
Days | 13.09 [2.87 to 27.04] | 13.1 [2.99 to 15.10]

7. Secondary Outcome: AUC 0-t (h*ng/mL)
Description: Area under the drug concentration (h*ng/mL) (AUC) vs time curve on Days 1 and 2
Time Frame: Pre- dose (within 30mins prior to each dose) and 1, 4 and 8 hours after each dose.
Population: Day 1 data only available for 7 subjects
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ANA001
Number analyzed (Participants) | 11
h*ng/mL
  Day 1: AUC 0-t (h*ng/mL): number analyzed (Participants) | 7
  Day 1: AUC 0-t (h*ng/mL) | 1728.6 (1410.21)
  Day 2: AUC 0-t (h*ng/mL) | 2839.0 (1702.25)

8. Secondary Outcome: Cmax (ng/mL)
Description: Maximum post dose plasma drug concentration on [Cmax (ng/mL)] Days 1 and 2
Time Frame: Pre- dose (within 30mins prior to each dose) and 1, 4 and 8 hours after each dose.
Population: Day 1 data only available for 7 subjects
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ANA001
Number analyzed (Participants) | 11
ng/mL
  Day 1: Cmax (ng/mL): number analyzed (Participants) | 7
  Day 1: Cmax (ng/mL) | 348.06 (212.343)
  Day 2: Cmax (ng/mL) | 435.91 (204.059)

9. Secondary Outcome: Tmax (h)
Description: Time to maximum post dose plasma drug concentration on [Tmax (h)] Days 1 and 2
Time Frame: Pre- dose (within 30mins prior to each dose) and 1, 4 and 8 hours after each dose.
Population: Day 1 data only available for 7 subjects
Measure: Mean (Standard Deviation); unit: (h)
Arm/Group | ANA001
Number analyzed (Participants) | 11
(h)
  Day 1: Tmax (h): number analyzed (Participants) | 7
  Day 1: Tmax (h) | 4.884 (2.3139)
  Day 2: Tmax (h) | 3.983 (2.4002)

ADVERSE EVENTS:
Time Frame: TEAEs are any adverse events that emerge on or after first dosing and up to 28 days after last dose during follow-up.
Arm/Group | ANA001 | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 2/22 | 3/23
Serious Adverse Events (participants affected / at risk) | 3/22 | 6/23
Other Adverse Events (participants affected / at risk) | 16/22 | 12/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANA001 (N=22) | Matching Placebo (N=23)
Septic shock (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANA001 (N=22) | Matching Placebo (N=23)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 5 (5)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Oral candiasis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediatinum (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increases (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 2 (2)
Fibrin D dimer increased (Investigations) | 0 (0) | 2 (2)
Granulocyte count increased (Investigations) | 0 (0) | 1 (1)
Immature granulocyte percentage increased (Investigations) | 0 (0) | 1 (1)
Klebsiella test positive (Investigations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT04603924/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT04603924/SAP_001.pdf